CLINICAL TRIAL: NCT01414972
Title: The Effect of Vitamin A Supplementation on Gene Expression of Cytokine Secreted by T CD4+ Lymphocyte in Atherosclerotic Patients
Brief Title: The Effect of Vitamin A on Atherosclerosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Ali Akbar Saboor Yaraghi /Assistant Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 89-01-27-10471
Record Dates: First submitted 2011-02-14; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Atherosclerosis
Keywords: Atherosclerosis; Coronary Artery Disease; Vitamin A; CD4-Positive T-Lymphocytes; gene expression
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease | interventions — Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- patients with atherosclerosis/ vitamin A (Active Comparator): patients with angiographically confirmed CAD (defined as luminal stenosis ≥50% in at least one major coronary artery branch)who receive 25000 IU/day vitamin A
  Interventions: Drug: Vitamin A
- patients with atherosclerosis/ placebo (Placebo Comparator): patients with angiographically confirmed CAD (defined as luminal stenosis ≥50% in at least one major coronary artery branch)who receive placebo
  Interventions: Drug: placebo
- people without athrosclerosis/ vitamin a (Active Comparator): people in whom significant (e.g. stenosis ≥ 50%) CAD is ruled out by coronary angiography, who receive 2500 Iu/day vitamin A
  Interventions: Drug: Vitamin A

INTERVENTIONS:
Drug: Vitamin A — 1 cap vitamin A 25000 IU/day for 3 month
  Arms: patients with atherosclerosis/ vitamin A; people without athrosclerosis/ vitamin a
Drug: placebo — 1 cap placebo/day for 3 month
  Arms: patients with atherosclerosis/ placebo

SUMMARY:
The aim of this study is the comparison between the effects of supplementation with 25000 IU preformed vitamin A (retinyl palmitate) or placebo for 4 months on gene expression of T CD4+ lymphocyte in atherosclerotic patients(documented with angiography).

DETAILED DESCRIPTION:
Atherosclerosis, the leading cause of death and disability in the world, is considered an inflammatory disease with a complex etiology. The immune system has a prominent role in the formation, development and destabilization of atherosclerotic plaques. A whole range of identified cytokines have been shown to play a part in atherogenesis, some with proatherogenic properties while others having antiatherogenic properties. With increasing evidence for the significant role of inflammation and the cytokines involved together with the Th1/Th2 imbalance in atherosclerosis and its progression to Coronary artery diseases (CADs), the control of cytokine production may become potential therapeutic targets and modulation of the Th1/Th2 balance may provide a new pharmacological tool to treat this disease. Vitamin A (VA) or VA-like analogs known as retinoids, are potent hormonal modifiers of type 1 or type 2 responses but a definitive description of their mechanism(s) of action is lacking. high level dietary vitamin A enhances Th2 cytokine production and IgA responses, and is likely to decrease Th1 cytokine production. Retinoic acid inhibits IL 12 production in activated macrophages, and RA pretreatment of macrophages reduces IFNγ production and increases IL4 production in antigen primed CD4 T cells. Supplemental treatment with vitamin A or retinoic acid (RA) decreases IFNγ and increases IL5, IL10, and IL4 production. Thus, vitamin A deficiency biases the immune response in a Th1 direction, whereas high level dietary vitamin A may bias the response in a Th2 direction.

ELIGIBILITY:
Inclusion Criteria:

• The criteria for enrollment of the patients and control subjects is consecutive patients of both sexes referred to the Division of Cardiology of the one of the Hospitals of Tehran University of Medical Sciences for coronary angiography for investigation of chest pain and/or suspected CAD.

Exclusion Criteria:

* Patients who have diseases which affect on Th1/Th2 balance such as asthma, active viral infections, and autoimmune diseases, OR
* Patients who have allergy to vitamin A compounds, OR
* Patients who have used vitamin supplements in last 3 months.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
serum Total cholesterol | Change from baseline at 4 months
serum HDL cholesterol | Change from baseline at 4 months
serum triglycerides level | Change from baseline at 4 months
RBP/ TTR ratio | Change from baseline at 4 months
PBMC's proliferation (BrdU colorimetric) | Change from baseline at 4 months
complete blood count (CBC) | Change from baseline at 4 months
SGOT | Change from baseline at 4 months
SGPT | Change from baseline at 4 months

SECONDARY OUTCOMES:
gene expression of T-bet, INF-gamma, IL-4, GATA3, IL-17, RORc, IL-10, FOXP3 (Relative quantification) | Change from baseline at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ali Akbar saboor Yaraghi, PhD, Study Chair — Tehran University of Medical Sciences; Azadeh Mottaghi, PhD student, Principal Investigator — Tehran University of Medical Siences
Locations (1):
- Tehran University of Medical Sciences, School of Public Health, Tehran, Iran